CLINICAL TRIAL: NCT06096376
Title: Predictors of High-Flow Nasal Cannula Failure (HFNC) in Patients With Acute Hypoxemic Respiratory Failure (AHRF) Using Diaphragm Ultrasound Parameters
Brief Title: Predictors of HFNC Failure in Patients With AHRF Using Diaphragm Ultrasound
Acronym: ULTRAFLOW
Status: Completed | Type: Observational
Sponsor: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Wincy Wing-Sze Ng, Associate Consultant, Adult Intensive Care Unit, Queen Mary Hospital, Hong Kong
Other Study IDs: UW 23-086-02
Record Dates: First submitted 2023-10-13; First posted 2023-10-23 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Acute Hypoxemic Respiratory Failure
Keywords: Acute Hypoxemic Respiratory Failure; High Flow Nasal Cannula; Diaphragm Ultrasound
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diaphragm Ultrasound — Diaphragm ultrasound to assess respiratory muscle function and respiratory efficiency

SUMMARY:
Ultrasound of the diaphragm is an easily reproducible bedside tool that provides a non-invasive measurement of inspiratory muscle function and respiratory efficiency. The diaphragmatic thickness correlates with the strength and muscle shortening and is reflective of its contribution to the respiratory workload. Diaphragm thickening fraction (DTF) has been shown to be predictive of extubation failure in ventilated patients. However, whether measurements of DTF are predictive of high flow nasal cannula (HFNC) outcomes in patients with acute hypoxemic respiratory failure (AHRF) remains unknown. The objective of this study is to identify predictors of HFNC failure by diaphragm ultrasound and to compare its performance with the well-established ROX index.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧ 18; AND
* Acute hypoxemic respiratory failure (AHRF), defined by respiratory rate of greater than 25 breaths per minute and a ratio of the PaO2 to the fraction of inspired oxygen (PaO2 / FiO2) of less than 300, and use of accessory muscles of respiration or paradoxical abdominal motion; AND
* Required ventilatory support with high-flow nasal cannula (HFNC)

Exclusion Criteria:

* Patients suffering from hypercapnic respiratory failure; OR
* AHRF secondary to conditions that are indicated for non-invasive ventilation (NIV) (e.g. acute exacerbation of COPD, cardiogenic pulmonary edema); OR
* Use of NIV or invasive mechanical ventilation (IMV) prior to HFNC initiation; OR
* Patients with imminent need for endotracheal intubation and invasive mechanical ventilation (IMV); OR
* Patients with known or suspected diaphragm paralysis; OR
* Pregnancy; OR
* Patients with abdominal compartment syndrome; OR
* Use of HFNC for more than 12 hours prior to ICU admission; OR
* Patients with suboptimal diaphragm ultrasound image quality for data processing; OR

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from acute hypoxemic respiratory requiring ventilatory support with high flow nasal cannula
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
High flow nasal cannula (HFNC) therapeutic failure | From the start of recruitment into study (i.e. start of HFNC use), till the date of study endpoint (i.e., step up to non-invasive ventilation, intubation, death on HFNC, or weaned off HFNC, whichever came first), assessed up to 4 weeks.
  Predictive value of diaphragm ultrasound in detecting high flow nasal cannula (HFNC)therapeutic failure in patients with acute hypoxemic respiratory failure (AHRF)

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided